CLINICAL TRIAL: NCT01989728
Title: Prevalence and Effect of Detecting Common Mental Disorders in Long-term Sickness Absence
Acronym: PRW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region MidtJylland Denmark (Other)
Responsible Party: Principal Investigator, Hans Joergen Soegaard, MD, consultant, prof. ph.d., Region MidtJylland Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sickness absence 1; RA (Other: Ringkøbing Amt)
Record Dates: First submitted 2013-11-08; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Psychiatric Disorders; Common Mental Disorders; Depression; Anxiety; Somatoform Disorder
Keywords: sickness absence, return to work, psychiatric examination, feedback, psychological distress, quality of life, attrition analysis, multiple imputation
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders; Somatoform Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- care as usual (Active Comparator)
  Interventions: Procedure: psychiatric examination and feedback
- psychiatric examination and feedback (Experimental)
  Interventions: Procedure: psychiatric examination and feedback

INTERVENTIONS:
Procedure: psychiatric examination and feedback

SUMMARY:
The hypothesis was that a large fraction of individuals with common mental disorders were undetected in long-term sickness and that detection of the disorders by screening, a psychiatric diagnostic examination and feedback to the individuals, primary care, and rehabilitation officers improved return to work, improved quality of life and reduced psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* First sick-listing between August 30, 2004 and August 29, 2005 in six municipalities (118,000 inhabitants)

Exclusion Criteria:

* Unable to understand Danish and absence due to pregnancy

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1121 (Actual)
Dates: Start 2004-11; Primary Completion 2005-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
duration until return to work | 1-2 years
  Included individuals were followed until payment of sickness absence compensation was ended

SECONDARY OUTCOMES:
Psychological distress by subscales of Hopkins Symptom Checklist Revised (SCL-90-R) | 1 year
  At baseline when entering long-term sickness absence (eight weeks of continuous sickness absence) the psychological distress was measured

OTHER OUTCOMES:
Quality of life by means of Social Functioning) SF-36 | 1 year
  At baseline when entering long-term sickness absence (eight weeks of continuous sickness absence) the quality of life was measured

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Research Unit west, regional Psychiatric Services West, Herning, Denmark

REFERENCES:
- [Result] Sogaard HJ, Bech P. Psychiatric disorders in long-term sickness absence -- a population-based cross-sectional study. Scand J Public Health. 2009 Sep;37(7):682-9. doi: 10.1177/1403494809344357. Epub 2009 Aug 21. PMID 19700479
- [Result] Sogaard HJ, Bech P. Psychometric analysis of common mental disorders -- Screening Questionnaire (CMD-SQ) in long-term sickness absence. Scand J Public Health. 2009 Nov;37(8):855-63. doi: 10.1177/1403494809344653. Epub 2009 Aug 28. PMID 19717571
- [Result] Sogaard HJ. Choosing screening instrument and cut-point on screening instruments. A comparison of methods. Scand J Public Health. 2009 Nov;37(8):872-80. doi: 10.1177/1403494809344442. Epub 2009 Aug 28. PMID 19717573
- [Result] Sogaard HJ, Bech P. The effect on length of sickness absence by recognition of undetected psychiatric disorder in long-term sickness absence. A randomized controlled trial. Scand J Public Health. 2009 Nov;37(8):864-71. doi: 10.1177/1403494809347551. Epub 2009 Sep 7. PMID 19736249
- [Result] Sogaard HJ, Bech P. Predictive validity of common mental disorders screening questionnaire as a screening instrument in long term sickness absence. Scand J Public Health. 2010 Jun;38(4):375-85. doi: 10.1177/1403494809350520. Epub 2009 Oct 22. PMID 19850649
- [Result] Sogaard HJ, Bech P. Compensating for non-response in a study estimating the incidence of mental disorders in long-term sickness absence by a two-phased design. Scand J Public Health. 2010 Aug;38(6):625-32. doi: 10.1177/1403494810373673. Epub 2010 Jun 7. PMID 20529969
- [Result] Sogaard HJ, Bech P. The effect of detecting undetected common mental disorders on psychological distress and quality of life in long-term sickness absence: a randomised controlled trial. Scand J Public Health. 2010 Dec;38(8):845-56. doi: 10.1177/1403494810379292. Epub 2010 Jul 22. PMID 20651000